CLINICAL TRIAL: NCT02762903
Title: Lesser Tuberosity Osteotomy Versus Tenotomy for Subscapularis Repair During Total Shoulder Arthroplasty
Brief Title: Lesser Tuberosity Osteotomy for Subscapularis Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAE1446
Record Dates: First submitted 2016-04-19; First posted 2016-05-05 (Estimated); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis
Keywords: Shoulder arthroplasty; Lesser Tuberosity Osteotomy; Subscapularis tenotomy
MeSH Terms: conditions — Osteoarthritis | interventions — theasinensin A; Shoulder Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tenotomy (Active Comparator): Subjects will receive shoulder prosthesis for subscapularis repair during TSA with tenotomy technique.
  Interventions: Procedure: TSA with tenotomy technique; Device: Shoulder prosthesis
- Osteotomy (Active Comparator): Subjects will receive shoulder prosthesis for subscapularis repair during TSA with lesser tuberosity osteotomy technique.
  Interventions: Procedure: TSA with lesser tuberosity osteotomy technique; Device: Shoulder prosthesis

INTERVENTIONS:
Procedure: TSA with tenotomy technique — Standard procedure: Utilization of tenotomy for mobilization of subscapularis during total shoulder arthroplasty (TSA). The subscapularis tendon is incised close to its attachment on the humerus. The Tendon is repaired with sutures.
  Arms: Tenotomy
Procedure: TSA with lesser tuberosity osteotomy technique — Standard procedure: Utilization of the osteotomy to mobilize the subscapularis during TSA. A small fleck of bone is removed from humerus, the subscapularis tendon is still attached. The fleck of bone is reattached with sutures.
  Arms: Osteotomy
Device: Shoulder prosthesis — Standard procedure: Total shoulder arthroplasty replaces both components of the "ball and socket" joint with a metal device.

SUMMARY:
The primary objective of this study is to assess the clinical effectiveness of two different techniques used for subscapularis tendon repair during total shoulder replacement. The investigators hypothesize that participants who receive a newer repair technique called a lesser tuberosity osteotomy will have lower rates of postoperative subscapularis muscle dysfunction and rupture as compared to those who receive the traditional tenotomy repair.

DETAILED DESCRIPTION:
The subscapularis tendon is mobilized during total shoulder arthroplasty in order to gain anterior access to the glenohumeral joint. Postoperative subscapularis dysfunction is being recognized more frequently and has been reported in >65% of patients following shoulder arthroplasty with a soft-tissue repair. Subscapularis dysfunction has been associated with poor functional outcomes including tendon rupture and anterior instability, a major indication for revision surgery. Recent studies suggest that a standard subscapularis tenotomy with primary tendon repair may lead to failure of the repair and decreased functional outcomes as compared to a more novel lesser tuberosity osteotomy technique. The investigators study aims to validate the results of the current literature in a prospective randomized controlled trial, which to their knowledge has not been reported on this topic.Investigators will compare clinical outcomes following these two techniques during total shoulder arthroplasty. Participants undergoing total shoulder replacement will be randomized to receive either a lesser tuberosity osteotomy or tenotomy with primary subscapularis tendon repair. All other procedures conducted in this study are considered standard of care except for ultrasounds, which are conducted for research purposes in the subscapularis tenotomy group. Postoperative outcomes will be monitored objectively and subjectively at routine postoperative office visits using physical exam, imaging (X-rays and ultrasounds), and questionnaires. If the hypothesis is proven to be true, the investigators will establish gold-standard evidence for the use of the newer osteotomy technique to improve patient satisfaction and mobility following shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients already scheduled for total shoulder arthroplasty

Exclusion Criteria:

* Unable to provide information throughout postoperative recovery and attend subsequent office visits thereafter (a minimum of one year).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William N. Levine, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Levine WN, Munoz J, Hsu S, Byram IR, Bigliani LU, Ahmad CS, Kongmalai P, Shillingford JN. Subscapularis tenotomy versus lesser tuberosity osteotomy during total shoulder arthroplasty for primary osteoarthritis: a prospective, randomized controlled trial. J Shoulder Elbow Surg. 2019 Mar;28(3):407-414. doi: 10.1016/j.jse.2018.11.057. PMID 30771825

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tenotomy | Osteotomy
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenotomy | Osteotomy | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Count of Participants; unit: Participants]
  0-18 years | 0 | 0 | 0
  At least 18 years old | 30 | 30 | 60
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex/gender were not collected from participants.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Radiologic Evidence of Anatomic Healing
Description: Tendon healing/tuberosity union based on radiographs
Time Frame: Post operative at 1 year
Population: Only includes participants who completed the final follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenotomy | Osteotomy
Number analyzed (Participants) | 30 | 29
Participants | 26 | 27

2. Secondary Outcome: Mean Visual Analogue Pain Scale (VAS)
Description: Pain indication measurement where 0 indicates no pain and 10 indicates worst possible pain. Mean score is reported without a range or standard deviation.
Time Frame: 1 year post-operatively
Population: Only includes participants who completed the final follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenotomy | Osteotomy
Number analyzed (Participants) | 30 | 29
score on a scale | 1.9 (NA) — The standard deviation was not calculated. Raw data existed during the study period of 2009 to 2013. This record was completed and published in 2016 without results. The data was subsequently destroyed because the data retention period had ended. This study closed with the IRB in 2017 and further analysis cannot be conducted. As of the current year, 2024, all the raw data for this study no longer exists. The standard deviation cannot be calculated without the raw data. | 1.8 (NA) — The standard deviation was not calculated. Raw data existed during the study period of 2009 to 2013. This record was completed and published in 2016 without results. The data was subsequently destroyed because the data retention period had ended. This study closed with the IRB in 2017 and further analysis cannot be conducted. As of the current year, 2024, all the raw data for this study no longer exists. The standard deviation cannot be calculated without the raw data.

3. Secondary Outcome: Forward Elevation (FE) Strength
Description: Strength testing with Dynamometer in forward elevation was conducted to determine the mean in FE strength.
Time Frame: 1 year post-operatively
Population: Only includes participants who completed the final follow-up.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Tenotomy | Osteotomy
Number analyzed (Participants) | 30 | 29
degrees | 153 (7) | 150 (6)

4. Secondary Outcome: Total Intra-Operative Time
Description: To be recorded in minutes, and documented by the surgical team
Time Frame: From incision time to time of complete skin closure
Population: Only includes participants who completed the final follow-up.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Tenotomy | Osteotomy
Number analyzed (Participants) | 30 | 29
minutes | 129.3 (NA) — The standard deviation was not calculated. Raw data existed during the study period of 2009 to 2013. This record was completed and published in 2016 without results. The data was subsequently destroyed because the data retention period had ended. This study closed with the IRB in 2017 and further analysis cannot be conducted. As of the current year, 2024, all the raw data for this study no longer exists. The standard deviation cannot be calculated without the raw data. | 152.7 (NA) — The standard deviation was not calculated. Raw data existed during the study period of 2009 to 2013. This record was completed and published in 2016 without results. The data was subsequently destroyed because the data retention period had ended. This study closed with the IRB in 2017 and further analysis cannot be conducted. As of the current year, 2024, all the raw data for this study no longer exists. The standard deviation cannot be calculated without the raw data.

5. Secondary Outcome: Total Subscapularis Repair Time (in Minutes)
Description: To be recorded in minutes, and documented by the surgical team
Time Frame: From glenoid implantation to completion of tendon or osteotomy repair
Population: Only includes participants who completed the final follow-up.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Tenotomy | Osteotomy
Number analyzed (Participants) | 30 | 29
minutes | 34.3 (NA) — The standard deviation was not calculated. Raw data existed during the study period of 2009 to 2013. This record was completed and published in 2016 without results. The data was subsequently destroyed because the data retention period had ended. This study closed with the IRB in 2017 and further analysis cannot be conducted. As of the current year, 2024, all the raw data for this study no longer exists. The standard deviation cannot be calculated without the raw data. | 39.3 (NA) — The standard deviation was not calculated. Raw data existed during the study period of 2009 to 2013. This record was completed and published in 2016 without results. The data was subsequently destroyed because the data retention period had ended. This study closed with the IRB in 2017 and further analysis cannot be conducted. As of the current year, 2024, all the raw data for this study no longer exists. The standard deviation cannot be calculated without the raw data.

6. Secondary Outcome: External Rotation (ER) Strength
Description: Strength testing with Dynamometer in external rotation.
Time Frame: 1 year post-operatively
Population: Only includes participants who completed the final follow-up.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Tenotomy | Osteotomy
Number analyzed (Participants) | 30 | 29
degrees | 50 (2) | 52 (3)

ADVERSE EVENTS:
Time Frame: Up to 1 year after surgery.
Arm/Group | Tenotomy | Osteotomy
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 5/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenotomy (N=30) | Osteotomy (N=30)
Tear of Supraspinatus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Partial-thickness, bursal-sided tear of the supraspinatus managed nonoperatively.
Subacromial impingement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subacromial impingement requiring arthroscopic bursectomy and anterior acromioplasty
Pain (General disorders) | 0 (0) | 1 (1) — Pain developed at 3 months postoperatively owing to a loose cerclage wire, requiring hardware removal and lysis of adhesions.
Transient post-operative radial nerve palsy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Subacromial bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Trapezius spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The standard deviation for Outcome Measure #2,4,5 was not calculated. Raw data existed during the study period of 2009 to 2013. This record was completed and published in 2016 without results. The data was subsequently destroyed because the data retention period had ended. This study closed with the IRB in 2017 and further analysis cannot be conducted. As of the current year, 2024, all the raw data for this study no longer exists. The standard deviation cannot be calculated without the raw data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes